CLINICAL TRIAL: NCT04304105
Title: Natural Progression of High-Risk Chronic Limb-Threatening Ischemia: The CLariTI Study
Status: Completed | Type: Observational
Sponsor: LimFlow, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: LF-CA-PR-8
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Critical Limb Ischemia; Peripheral Artery Disease
Keywords: CLI
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this observational registry is to track the clinical progression of chronic limb-threatening ischemia (CLTI) and incidence of death, amputation, and revascularization attempts over a one-year period.

DETAILED DESCRIPTION:
The objective of this observational registry is to track the clinical progression of chronic limb-threatening ischemia (CLTI) and incidence of death, amputation, and revascularization attempts over a one-year period.

The study population is comprised of Rutherford 5 and 6 CLTI subjects who have hemodynamic evidence of severely diminished arterial inflow of a peripheral limb and:

1. 2 revascularizations in the last 6 months that failed to resolve symptoms, OR
2. have inadequate popliteal, tibial, or pedal revascularization target

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be ≥18 years of age
2. Subject is Rutherford 5 or 6 classification with hemodynamic evidence of severely diminished arterial inflow of a peripheral limb and: a) 2 revascularizations in the last 6 months that failed to resolve symptoms, OR b) An inadequate popliteal, tibial, or pedal revascularization target
3. Subject is willing and able to sign the informed consent form and willing to participate in the phone follow-ups.

Exclusion Criteria:

1. Any significant concurrent psychological or social condition (e.g., no support person/network), which may significantly interfere with the subject's optimal participation in the study, in the opinion of the investigator.
2. Subject is participating in the PROMISE II Clinical Trial.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population is comprised of Rutherford 5 and 6 CLTI subjects who have hemodynamic evidence of severely diminished arterial inflow of a peripheral limb and:
  1. 2 revascularizations in the last 6 months that failed to resolve symptoms, OR
  2. have inadequate popliteal, tibial, or pedal revascularization target
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-09-12 (Actual)

PRIMARY OUTCOMES:
Amputation Free Survival (AFS) | 12 months
  Defined as freedom from major (above ankle) amputation and death

SECONDARY OUTCOMES:
Minor Amputation | 12 months
  Number of patients with below-ankle amputation of the index limb
Change in Rutherford Classification | 6 months and 12 months
  Defined as a change of one class or greater, as evaluated at 6 and 12 months

CONTACTS AND LOCATIONS:
Locations (25):
- United States (24):
  - LA Foot & Ankle Clinic - St. Vincent's Hospital, Los Angeles, California
  - Harbor- UCLA Medical Center, Torrance, California
  - Denver Veterans Affairs Medical Center, Denver, Colorado
  - The Cardiac and Vascular Institute, Gainesville, Florida
  - Unity Point Health, Des Moines, Iowa
  - Ochsner Medical Center, Kenner, Louisiana
  - MedStar D.C., Hyattsville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Ascension St. John Detroit, Detroit, Michigan
  - St. Lukes Mid America, Kansas City, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - APCNC (Wake Med), Cary, North Carolina
  - East Carolina University (ECU, Vidant Medical), Greenville, North Carolina
  - Coastal Carolina Surgical, Wilmington, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Anderson Heart and Vascular, Anderson, South Carolina
  - Coastal Vascular and Vein Center, Charleston, South Carolina
  - Prisma Health, Greenville, South Carolina
  - Seton Heart Institute, Austin, Texas
  - Austin Radiological Association, Austin, Texas
  - Baylor College of Medicine, Houston, Texas
  - UT-San Antonio, San Antonio, Texas
  - VCU, Virginia Commonwealth University Health System, Richmond, Virginia
- San Lucas Hospital, Ponce, Puerto Rico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Powell RJ, Mullin CM, Clair DG, Shishehbor MH, Dua A. Comparison of Transcatheter Arterialization of Deep Veins to Standard of Care in Patients with No-Option Chronic Limb Threatening Ischemia. Ann Vasc Surg. 2024 Feb;99:50-57. doi: 10.1016/j.avsg.2023.08.010. Epub 2023 Oct 18. PMID 37858666